CLINICAL TRIAL: NCT00000354
Title: Safety Evaluation of Lofexidine for Treatment of Opioid Withdrawal
Brief Title: Evaluation of Lofexidine for Treatment of Opioid Withdrawal - 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Purpose: Treatment
Other Study IDs: NIDA-3-0012-3; Y01-3-0012-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1996-07

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — lofexidine

INTERVENTIONS:
Drug: Lofexidine

SUMMARY:
The purpose of this study is to determine the safety of lofexidine in the treatment of opiate withdrawal. Preliminary data will also be obtained to assess the ability of lofexidine to alleviate opiate withdrawal signs and symptoms.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-07; Primary Completion 1997-09 (Actual); Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — PDVAMC Treatment Research Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States